CLINICAL TRIAL: NCT04493879
Title: Efficacy of Bioptron Light Therapy (BLT) on Post Chemotherapy Oral Mucositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Eid, assistant professor of physical therapy for surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 68
Record Dates: First submitted 2020-07-16; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Oral Mucositis (Ulcerative)
MeSH Terms: conditions — Stomatitis; Ulcer

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bioptron Light Therapy (BLT) group (Experimental): Received Bioptron Light Therapy (BLT) ten minutes every day for one month plus the routine medical treatment of oral mucositis(Analgesics, anti-inflammatory medication and antimicrobial therapy for any new mouth infections
  Interventions: Other: Bioptron Light Therapy (BLT)
- Routine medical care group (Experimental): Received only the routine medical care of oral mucositis for one month this consists of analgesics, anti-inflammatory treatment, and antimicrobial treatment for any new mouth infections
  Interventions: Other: Bioptron Light Therapy (BLT)

INTERVENTIONS:
Other: Bioptron Light Therapy (BLT) — BLT for 30 days 10 minutes every day. The treatment points displayed were: one point in the right jugal mucosa, one point in the left jugal mucosa, one point in the lower lip 's inner mucosa, analgesics, anti-inflammatory treatment, and antimicrobial treatment for any new mouth infections)

SUMMARY:
The study aimed to study the effect of Bioptron light therapy (BLT) on oral mucositis after receiving chemotherapy in patients with head and neck cancer,Oral mucositis (OM) is a common and severe acute side-effect of many oncologic treatments, especially in patients treated for head and neck cancer. It affects quality of life and require supportive care and proper treatment plane.

This study had been conducted on thirty cancer patients (head &neck) receiving chemotherapy & radiotherapy (males and females) with oral mucositis with ulceration and pain(grade 2 and more), their age ranged from 35 to 55 years, capable of understanding the study assessment method and willing to complete the current study, they were free from any immunodeficiency disorders or diseases that could impair the healing process and impact the results as diabetes mellitus. Patients were randomly allocated from patients from the National Cancer Institute, Cairo University. Group A (BLT group): This group consisted of 15 patients receiving BLT for about 10 minutes every day for thirty days in addition to routine oral mucositis medical care (Analgesics, anti-inflammatory treatment and antimicrobial treatment for any new mouth infections), Group B (Control group): This group consisted of 15 patients receiving daily routine oral mucositis medical care(Analgesics, anti-inflammatory treatment and antimicrobial treatment for any new mouth infections) for thirty days The methods of evaluation in the current study were the WHO oral mucositis scale (OMS) and the Common toxicity criteria scale (CTCS). At the same time, the treatment equipment was the polarized light therapy device Bioptron Compact III (PAG-860 manufactured in Switzerland) Assessment by WHO oral mucositis scale and (OMS) and (CTCS) were used before treatment and after treatment to measure improvement in oral mucositis.

The results of WHO oral mucositis scale (OMS) and the Common toxicity criteria scale (CTCS) were assessed first at the beginning of the study and one month after the end of the study; calculation of mean, standard deviation, minimum and maximum for each group was done by descriptive statistics, means comparison between the two groups pre and post-application and within each group was made using The t-test. With a level of significance Alpha point of 0.05

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients (head &neck) receiving chemotherapy & radiotherapy
* Males and females
* Age ranged from 35-55 years
* All patients capable of understanding the study assessment method and willing to complete the current study
* Patients free from any immunodeficiency disorders or diseases that could impair the healing process and impact the results as diabetes .

Exclusion Criteria:

* Patients suffering from immunodeficiency disorders or diseases that could impair the healing process and impact the results as diabetes .
* Cognitive impairment

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Oral Ulceration | 30 days
  WHO oral mucositis scale (OMS) and the Common toxicity criteria scale (CTCS)

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Eid, Principal Investigator — Ass.Prof
Locations (1):
- Marwa Eid, Cairo, Egypt